CLINICAL TRIAL: NCT06461923
Title: Development and Feasibility Study of the Home-based Gait Rehabilitation Service by Using the Insole-type Gait Analysis Device for Children With Cerebral Palsy
Brief Title: Home-based Gait Rehabilitation Service Using the Insole-type Gait Analysis Device for Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 4-2023-1407
Record Dates: First submitted 2024-05-28; First posted 2024-06-17 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Gait Disorders, Neurologic; Cerebral Palsy
Keywords: gait parameters; smart insole; home-based exercise; monitoring system; rehabilitation
MeSH Terms: conditions — Gait Disorders, Neurologic; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insole wearing (Experimental)
  Interventions: Device: Insole wearing

INTERVENTIONS:
Device: Insole wearing — The insole-wearing group is instructed to wear the insole gait analysis device as frequently and for as long as possible during outdoor activities. Participants receive feedback during 3rd to 4th week via telephone. Following a period of 6 weeks, an evaluation of the usability and satisfaction of the insole gait analysis device will be conducted.

SUMMARY:
Walking is a crucial daily activity that requires complex coordination of muscular systems. It is essential for bone and muscle health, cardiovascular fitness, and activities of daily living, making it an important indicator of prognosis and patient function. Insole gait analysis devices are affordable and easy to use, and they align well with standardized 3D gait analysis. However, their use outside of hospital settings is limited.

This study aims to assess the usability and satisfaction of utilizing insole gait analysis devices for monitoring and providing feedback on the walking status of children with cerebral palsy exhibiting walking impairments in a home environment. Additionally, adherence to a home-based exercise program developed in this study will be evaluated.

DETAILED DESCRIPTION:
The screening test is conducted after obtaining consent, and it involves assessing whether the subject can independently walk more than 10 meters, regardless of the use of assistive devices, following an evaluation of their baseline symptoms and signs.

Subjects who pass the screening test are provided with information about their current walking status and what constitutes normal walking. Following the initial evaluation, they are instructed to participate in the 6-week home exercise program and how to record an exercise log. Additionally, researchers provide participants with an insole gait analysis device and instruct them on its operation, encouraging prolonged usage to ensure that usage time and walking patterns are recorded.

Based on the collected measurement data, feedback is provided over the phone at weeks 3 to 4. After completing the 6-week home exercise program, a final evaluation is conducted in the same manner as the initial evaluation. Satisfaction with the insole gait analysis device is assessed only at the time of the final evaluation.

Usage and satisfaction with the insole gait analysis device will be analyzed, and evaluation indicators will be compared before and after the home exercise program. Additionally, adherence to the home exercise program will be evaluated through exercise logs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with cerebral palsy aged 7 to 18 years old
2. Patients classified as Gross Motor Function Classification System level 1 or 2
3. Individuals who visited Severance Hospital, comprehended the study, agreed to participate, and submitted the informed consent form

Exclusion Criteria:

1. Individuals with complications such as severe foot deformities where the sensors of the insole gait analysis device cannot be recognized
2. In addition to above, individuals with clinically significant findings deemed inappropriate for this study by the study director or person in charge based on medical judgment

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
6-minute Walking Test | This test results will be assessed two times: baseline and after 6 weeks

SECONDARY OUTCOMES:
Appendicular muscle mass (kg) | This test results will be assessed two times: baseline and after 6 weeks
  This outcome will be measured using bioelectrical impedance.
Height (cm) | This test results will be assessed two times: baseline and after 6 weeks
  This outcome will be measured using bioelectrical impedance.
Weight (kg) | This test results will be assessed two times: baseline and after 6 weeks
  This outcome will be measured using bioelectrical impedance.
Grip Strength Test (kg) | This test results will be assessed two times: baseline and after 6 weeks
The number of steps (n) | This test results will be assessed two times: baseline and after 6 weeks
  This outcome will be collected using an insole-type gait analyzer.
Calories burned (kcal) | This test results will be assessed two times: baseline and after 6 weeks
  This outcome will be collected using an insole-type gait analyzer.
Activity time (min) | This test results will be assessed two times: baseline and after 6 weeks
  This outcome will be collected using an insole-type gait analyzer.
Activity distance (km) | This test results will be assessed two times: baseline and after 6 weeks
  This outcome will be collected using an insole-type gait analyzer.
Walking speed (m/s) | This test results will be assessed two times: baseline and after 6 weeks
  This outcome will be collected using an insole-type gait analyzer.
Stride length (cm) | This test results will be assessed two times: baseline and after 6 weeks
  This outcome will be collected using an insole-type gait analyzer.
Left-right gait balance (%) | This test results will be assessed two times: baseline and after 6 weeks
  This outcome will be collected using an insole-type gait analyzer.
10-meter Walking Test (m/s) | This test results will be assessed two times: baseline and after 6 weeks
Pediatric Balance Scale (scores) | This test results will be assessed two times: baseline and after 6 weeks
  The minimum score is 0 points, and the maximum score is 56 points. A higher score indicates better balance ability in children and a greater capacity to perform daily activities independently.
Gross Motor Function Classification System (levels) | This test results will be assessed two times: baseline and after 6 weeks
Korean version of Cerebral Palsy Quality of Life (scores) | This test results will be assessed two times: baseline and after 6 weeks
  If the participant is aged 8 or younger, the relevant questionnaire will be administered; otherwise, the Korean version of KIDSCREEN-52 will be used.
  The minimum score is 0 points, and the maximum score is 100 points. A higher score indicates a higher quality of life.
Korean version of KIDSCREEN-52 (Children & Adolescents) (scores) | This test results will be assessed two times: baseline and after 6 weeks
  If the participant is aged over 8, the relevant questionnaire will be administered.
  The minimum score is 52 points, and the maximum score is 260 points. A higher score indicates a higher quality of life.
Korean version of KIDSCREEN-52 (Parents) (scores) | This test results will be assessed two times: baseline and after 6 weeks
  The minimum score is 52 points, and the maximum score is 260 points. A higher score indicates a higher quality of life.
Satisfaction Survey for the Device (scores) | This test results will be assessed once: after 6 weeks
  The minimum score is 12, and the maximum score is 84 points. A higher score indicates lower satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Na Young Kim, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salzman B. Gait and balance disorders in older adults. Am Fam Physician. 2010 Jul 1;82(1):61-8. PMID 20590073
- [Result] Fritz S, Lusardi M. White paper: "walking speed: the sixth vital sign". J Geriatr Phys Ther. 2009;32(2):46-9. No abstract available. PMID 20039582
- [Result] Middleton A, Fritz SL, Lusardi M. Walking speed: the functional vital sign. J Aging Phys Act. 2015 Apr;23(2):314-22. doi: 10.1123/japa.2013-0236. Epub 2014 May 2. PMID 24812254
- [Result] Stolze H, Klebe S, Baecker C, Zechlin C, Friege L, Pohle S, Deuschl G. Prevalence of gait disorders in hospitalized neurological patients. Mov Disord. 2005 Jan;20(1):89-94. doi: 10.1002/mds.20266. PMID 15390043
- [Result] Giladi N, Horak FB, Hausdorff JM. Classification of gait disturbances: distinguishing between continuous and episodic changes. Mov Disord. 2013 Sep 15;28(11):1469-73. doi: 10.1002/mds.25672. PMID 24132835
- [Result] Carlon SL, Taylor NF, Dodd KJ, Shields N. Differences in habitual physical activity levels of young people with cerebral palsy and their typically developing peers: a systematic review. Disabil Rehabil. 2013 Apr;35(8):647-55. doi: 10.3109/09638288.2012.715721. Epub 2012 Oct 17. PMID 23072296
- [Result] Waltersson L, Rodby-Bousquet E. Physical Activity in Adolescents and Young Adults with Cerebral Palsy. Biomed Res Int. 2017;2017:8080473. doi: 10.1155/2017/8080473. Epub 2017 Dec 20. PMID 29423412
- [Result] O'Connell NE, Smith KJ, Peterson MD, Ryan N, Liverani S, Anokye N, Victor C, Ryan JM. Incidence of osteoarthritis, osteoporosis and inflammatory musculoskeletal diseases in adults with cerebral palsy: A population-based cohort study. Bone. 2019 Aug;125:30-35. doi: 10.1016/j.bone.2019.05.007. Epub 2019 May 8. PMID 31075418
- [Result] Mcphee PG, Claridge EA, Noorduyn SG, Gorter JW. Cardiovascular disease and related risk factors in adults with cerebral palsy: a systematic review. Dev Med Child Neurol. 2019 Aug;61(8):915-923. doi: 10.1111/dmcn.14028. Epub 2018 Sep 17. PMID 30221763
- [Result] Bulekbayeva S, Daribayev Z, Ospanova S, Vento S. Cerebral palsy: a multidisciplinary, integrated approach is essential. Lancet Glob Health. 2017 Apr;5(4):e401. doi: 10.1016/S2214-109X(17)30082-7. No abstract available. PMID 28288745
- [Result] Muro-de-la-Herran A, Garcia-Zapirain B, Mendez-Zorrilla A. Gait analysis methods: an overview of wearable and non-wearable systems, highlighting clinical applications. Sensors (Basel). 2014 Feb 19;14(2):3362-94. doi: 10.3390/s140203362. PMID 24556672
- [Result] Ngueleu AM, Blanchette AK, Maltais D, Moffet H, McFadyen BJ, Bouyer L, Batcho CS. Validity of Instrumented Insoles for Step Counting, Posture and Activity Recognition: A Systematic Review. Sensors (Basel). 2019 May 28;19(11):2438. doi: 10.3390/s19112438. PMID 31141973
- [Result] Andreoli A, Garaci F, Cafarelli FP, Guglielmi G. Body composition in clinical practice. Eur J Radiol. 2016 Aug;85(8):1461-8. doi: 10.1016/j.ejrad.2016.02.005. Epub 2016 Feb 15. PMID 26971404
- [Result] Lee SY. Handgrip Strength: An Irreplaceable Indicator of Muscle Function. Ann Rehabil Med. 2021 Jun;45(3):167-169. doi: 10.5535/arm.21106. Epub 2021 Jun 30. No abstract available. PMID 34233405
- [Result] Chrysagis N, Skordilis EK, Koutsouki D. Validity and clinical utility of functional assessments in children with cerebral palsy. Arch Phys Med Rehabil. 2014 Feb;95(2):369-74. doi: 10.1016/j.apmr.2013.10.025. Epub 2013 Nov 12. PMID 24239880

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT06461923/Prot_SAP_001.pdf